CLINICAL TRIAL: NCT02445547
Title: Umbilical Cord Mesenchymal Stem Cell Treatment for Crohn's Disease: A Randomized Controlled Clinical Trial
Brief Title: Umbilical Cord Mesenchymal Stem Cell Treatment for Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Collaborators: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCMSC-CD
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UC-MSCs (Experimental): UC-MSCs by peripheral intravenous infusion
  Interventions: Other: UC-MSCs by peripheral intravenous infusion
- control (Active Comparator): received hormone maintenance therapy
  Interventions: Drug: received hormone maintenance therapy

INTERVENTIONS:
Other: UC-MSCs by peripheral intravenous infusion
  Arms: UC-MSCs
Drug: received hormone maintenance therapy
  Arms: control

SUMMARY:
Stem cell transplantation has emerged as a relatively popular treatment that can help to regulate immunity, repair injury, and control inflammation. Several studies have used autologous stem cells or adipose-derived stem cells to treat Crohn's disease and its associated complications, and have achieved good efficacy. Thus far, the use of umbilical cord mesenchymal stem cells (UC-MSCs) to treat Crohn's disease has rarely been reported. In this study, UC-MSCs were used to treat patients with hormone-controlled Crohn's disease. We observed the disease control conditions, corticosteroid dosage changes, and treatment-related adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* moderate to severe Crohn's disease (Crohn's disease activity index (CDAI) between 220 and 450)
* had received hormone maintenance therapy for more than 6 months

Exclusion Criteria:

* active tuberculosis
* malignancy
* HIV
* syphilis
* hepatitis B
* hepatitis C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Crohn's disease activity index | 12 months

SECONDARY OUTCOMES:
Harvey-Bradshaw index | 12 months
Corticosteroid dosage | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shaanxi Provincial People's Hospital, XI Ail, Shaanxi, China